CLINICAL TRIAL: NCT02768831
Title: Minimal Occlusive Pressure With Cuffed ETTs: A Comparison of Two Different Techniques to Ensure a Tracheal Seal
Brief Title: ETT Cuff Leak: TV Ratios
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Senthil G. Krishna, Assistant Professor, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB16-00222
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Surgical Procedures, Operative
MeSH Terms: interventions — Tidal Volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cuffed ETT (Experimental)
  Interventions: Other: CPAP; Other: Tidal volume

INTERVENTIONS:
Other: CPAP — Sealing the airway by holding CPAP of 20 cmH2O in the anesthesia circuit and slowly inflating the cuff until no air leak is heard with a stethoscope placed in the suprasternal notch.
Other: Tidal volume — The ratio of the inspired to expired tidal volume will be determined using the following formula: (TVinspired - TV¬expired)/TVinspired. The peak inflating pressure (PIP) required to achieve the set TV will be noted. The air in the cuff will then be increased or decreased as needed to achieve a set delivered ratio of 0.9-1.0.
  Other Names: TV

SUMMARY:
In the past 5 years cuffed endotracheal tubes (ETT) have become the standard of care in pediatrics. However, hyperinflation of the cuff can compromise the tracheal mucosal perfusion while an inadequate seal may impact ventilation and potentially increase the risk of aspiration. Hence, the goal after placement of a cuffed ETT is to create a safe and effective tracheal seal. The two ways to measure that are to hold CPAP while listening for an audible leak and measuring the difference between the inspired and expired tidal volumes (TV). This is a prospective study to compare these two methods used to create a tracheal seal and measure the intracuff pressure after a satisfactory tracheal seal is established.

ELIGIBILITY:
Inclusion Criteria:

* Children who are scheduled to undergo GA with a cuffed ETT in place.

Exclusion Criteria:

* Any children with pre-existing tracheal/bronchial anomalies, patients with Down syndrome, patients with C-spine issues.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Intracuff pressure | Immediately following intubation
  Difference in intracuff pressure measured after inflation with CPAP and inflation with TV.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Moon K, Kitio SAY, Rice-Weimer J, Tobias JD. Regulation of Intracuff Pressure by Measurement of the Ratio of Expiratory to Inspiratory Tidal Volumes. Paediatr Anaesth. 2025 Nov;35(11):940-945. doi: 10.1111/pan.70045. Epub 2025 Sep 5. PMID 40913357